CLINICAL TRIAL: NCT01770210
Title: A Multicenter, Open-label, 30-week Observational Clinical Study to Examine the Progress of Patients After Leaving the Cardiology Clinic or Unit Due to Acute Cardiovascular Event.
Brief Title: Ekvasis of Atorvastatin (Antorcin®) Treatment in Patients With Acute Cardiovascular Events
Acronym: EKVASIS
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012-ATR-EL-34
Record Dates: First submitted 2013-01-14; First posted 2013-01-17 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Cardiovascular Disorders
Keywords: hypercholesterolemia; atorvastatin; cardiovascular events
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiovascular events: Patients on atorvastatin treatment hospitalised due to cardiovascular events
  Interventions: Drug: Patients on atorvastatin treatment

INTERVENTIONS:
Drug: Patients on atorvastatin treatment — Statins Therapy

SUMMARY:
In western societies hypercholesterolemia is one of the major and independent factors that predispose to cardiovascular disease and death from them. According to the clinical study ATTICA, conducted during the years 2001-2002, in which randomized 1514 men and 1528 women, rates of hypercholesterolemia observed in a sample of urban population was 39% for men and 37% women . The prevalence in the corresponding U.S. epidemiological study NIANES was 52% for men and 49% women. The relationship between cholesterol, lipid-lowering therapy and risk of cardiovascular disease appears to be quite clear in the secondary prevention trials, the 4S (Scandinavian Simvastatin Survival Study), CARE (Cholesterol And Recurrent Events) and LIPID (Long-term Intervention with Pravastatin in Ischemic Disease) which showed the benefits of lowering LDL cholesterol in patients with coronary artery disease. Despite these remarkable results, studies were secondary prevention as a major shortcoming, the lack of patients with acute coronary events. This gap came to cover the study MIRACL (Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering). In MIRACL study , atorvastatin 80 mg was evaluated in 3,086 patients (atorvastatin n = 1.538, placebo n = 1.548), acute coronary syndrome (myocardial infarction without Q-wave or unstable angina). Treatment was initiated during the acute phase after hospital admission and lasted for a period of 16 weeks. Treatment with atorvastatin 80 mg / day increased the latency of the combined primary endpoint, defined as death from any cause, nonfatal myocardial infarction, resuscitated cardiac arrest, or angina with objective evidence of myocardial ischemia requiring admission to hospital, indicating a risk reduction of 16% (p = 0,048). This was mainly due to a 26% reduction in re-hospitalization for angina with objective evidence of myocardial ischemia. The other secondary endpoints were not statistically significant by themselves (total: placebo: 22.2%, Atorvastatin: 22.4%).

Statins by reducing coronary syndromes, it appears that contribute to reducing the incidence of cardiovascular diseases. This is exactly what was observed in 4S, in which the incidence of chronic heart failure (CHF) during follow-up was 10.3% for those who received placebo and 8.3% in the simvastatin group, a finding which translates 19% reduction in heart failure (P <0,015) nationwide with the appearance episode (event) CV.

DETAILED DESCRIPTION:
Determination of cardiovascular risk

If the assessment of cardiovascular risk remains incomplete, can identify indicators that measure risk:

1. Framingham Risk Score: Includes age, sex, total and HDL-CHOL, and levels of blood pressure (can underestimate the risk in some patients).
2. PROCAM Risk Score: also includes triglycerides, fasting glucose tolerance and family history.
3. Reynolds Risk Score: Includes family history and levels of hsCRP.
4. Greek Score (www.hearts.org / greece). People with low risk The Framingham Risk Score shows <10% chance of cardiovascular disease over the next 10 years. Dealing mainly with healthy dietary intervention or drugs when the levels of LDL-CHOL> 190 mg / dL or atherogenic index (T-CHOL/HDL-CHOL)> 6.

Medication is necessary in individuals with familial hypercholesterolemia to reduce the LDL CHOL <100 mg / dL. For this reason, a careful family history taking physical examination. The Reynolds Risk Score may reclassify their low-risk patients at higher risk individuals.

Persons moderate risk This group includes mostly middle-aged people. The Framingham Risk Score shows 10-19% chance of cardiovascular disease over the next 10 years. However, a positive family history and high hsCRP (if available) can modify the level of risk. These people need to change my lifestyle for 3 months, but may then be necessary pharmacological lipid-lowering therapy in people with at least two major risk factors and levels of LDL-CHOL> 130 mg / dL. The administration of lipid-lowering therapy in people with levels of LDL-CHOL 100-129 mg / dL is recommended for people with multiple cardiometabolic risk factors (visceral obesity, prediabetes, hypertension, etc.). The increase of atheromatic index (> 5) and the presence of high (> 2 mg / L) levels of CRP (if available) are also indications for lipid lowering regardless of the levels of LDL-CHOL.

Major risk factors: age> 45 years (men),> 55 years (women), positive family history of premature cardiovascular disease [in the presence of major vascular events in first degree relatives <55 years (men), <65 years (women)], hypertension , HDL-CHOL <40 mg / dL, smoking.

Individuals at high risk The Framingham Risk Score shows> 20% chance of cardiovascular disease over the next 10 years. At-risk individuals include:

A. Individuals with documented atherosclerotic disease (coronary artery disease, stroke, a significant degree of carotid stenosis, peripheral arterial disease, intermittent claudication, or aneurysm of the abdominal aorta).

B. All type II diabetic patients and patients with type I diabetes individuals older than 40 years.

C. People with chronic kidney disease with glomerular filtration (GFR) <60 mL/min/1, 73 m2.

In these individuals need intensive lifestyle modification and direct administration lipid lowering medication such as statins.

According to the above that one epidemiological study nature that has the purpose of observing and recording the progress of patients after their exit from a cardiology clinic or hospital unit because the acid after a cardiovascular event has clinical relevance. Compliance with medical instructions, achieving treatment goals for lipids by the addition of atorvastatin and personalized medicine practice are open field study. So this will be the subject of this study in order to highlight the clinical significance of atorvastatin in achieving the objectives of lipids (mainly LDL-CHOL) in blood plasma of "sensitive" of this group of patients in the Greek population, as possible representative (qualitatively and quantitatively)sample.

Dyslipidemia

The lipids of the human body is cholesterol (useful for the synthesis of cell membranes, hormones adrenal and gonads, and is a component of bile, the liver secretes) and triglycerides (serve as fuel and energy storage in adipose tissue ). The dyslipidemias are disorders (quantitative or qualitative) of the metabolism of lipoprotein particles (LDL, chylomicrons, HDL, VLDL) that transport lipids in the body.

Categories dyslipidemias - Primary dyslipidemias

The most significant primary lipid disorders are:

1. Chylomicronemia (congenital or acquired): ↑ TRG → risk of acute pancreatitis.
2. Familial Hypercholesterolemia a Homozygous (1/1.000.000 people): ↑ LDL CHOL b heterozygous (1/500 people): ↑ LDL CHOL.
3. Mixed hyperlipidaemia Familial mixed (1/300 people): ↑ LDL-CHOL, ↑ TRG, ↓ HDL-CHOL.
4. Familial hypertriglyceridemia (1/2.000 people): ↑ TRG.
5. Familial decrease in HDL CHOL: ↓ HDL CHOL. Typically in patients with primary dyslipidemia needed medication. - Secondary dyslipidemias

In patients with abnormal lipid parameters of must exclude secondary dyslipidemias, ie disorders of lipid metabolism caused by diseases or drugs:

1. Diabetes
2. Hypothyroidism
3. Obstructive liver disease
4. Chronic kidney disease nephrotic syndrome-
5. Obesity
6. Alcohol abuse
7. Medications that cause dyslipidemia a progestin b Anabolic Steroids c Corticosteroids D. Diuretics in large doses e b-blockers f Antiretroviral Drugs Interferon g h. Retinoids Estrogen i tamoxifen. In patients with secondary dyslipidemia required treatment of primary disease. Determination cohort for screening (Table 1)

   * Men over 40 and post-menopausal women
   * People with atherosclerotic disease regardless of age or clinical findings suggestive of dyslipidemia
   * Patients with diabetes regardless of age
   * Patients with chronic kidney disease (eGFR <60 mL/min/1, 73 m2 or the presence of albuminuria)
   * People with a family history of premature coronary heart disease
   * People with hypertension
   * People with chronic inflammatory diseases (lupus erythematosus, rheumatoid arthritis, psoriasis or acquired immunodeficiency syndrome)
   * Adults who smoke
   * adult with sexual dysfunction
   * Overweight and obese subjects with BMI> 27 kg/m2
   * Relatives of people with inherited lipid disorders
   * Children with a family history of hyperlipidemia or cardiovascular disease or other risk factors.

Statins - Atorvastatin

The cornerstone of treatment of dyslipidemia are statins.

Before initiation of lipid lowering requires the identification of lipid parameters {total cholesterol, triglycerides, HDL cholesterol and calculated LDL cholesterol [from the equation LDL-CHOL = total cholesterol - (triglycerides / 5 + HDL cholesterol)]} after fasting 12 - 14 hours, while the determination of glucose levels of TSH (to exclude underlying hypothyroidism) and transaminases (AST / ALT) and CPK to control the undesirable effects. Repeat determination of these parameters in patients who achieved their goals of treatment 2 times a year or when changing the therapeutic regimen. Repeat laboratory tests (lipid control effectiveness and liver enzymes and CPK for security control) after 12 weeks: a reason to discontinue treatment if ALT> 3 times the upper normal range or CPK> 5 times the upper normal range or in patients with myalgias. It should be noted that not necessitate interruption of treatment with statins or deferral of treatment in individuals with small increases in transaminases or CPK, while in these patients should be seeking other underlying causes of elevated liver and muscle enzymes. The choice of drug and dosage depend on the percentage change in HDL-CHOL necessary to achieve the objectives. Statins are usually the evening before bedtime the night. The lipid-lowering therapy is therapy for life, and most importantly, the patient adherence to treatment. It should be noted that doubling the dose of a statin results in additional reduction of HDL-CHOL (LDL) cholesterol by 6%.

The main goal of treatment is to reduce HDL-CHOL

The non HDL-CHOL (= T-CHOL - HDL-CHOL), proposed as a secondary target of lipid lowering mainly in people with high triglycerides. The target for the non HDL-CHOL is 30 mg / dL higher than the target for the HDL-CHOL. The decrease in triglycerides (<150 mg / dL) and increased HDL-CHOL (> 40 mg / dL for men and> 50 mg / dL for women) is considered desirable targets mainly lipid lowering in diabetic patients and in patients with cardiometabolic risk factors. Has also been suggested as a target of treatment to reduce the atheromatous index (T-CHOL/HDL-CHOL <4).

Atorvastatin is indicated as an adjunct to diet to reduce elevated total cholesterol, LDL-cholesterol, apolipoprotein B and triglycerides in adults, adolescents and children aged 10 years and older with primary hypercholesterolaemia, including heterozygous familial hypercholesterolaemia combined (mixed) hyperlipidemia (type IIa and IIv by Fredrickson), when response to diet and other nonpharmacological measures is inadequate.

Atorvastatin is also indicated to reduce total cholesterol and LDL - cholesterol in adults with homozygous familial hypercholesterolemia as an adjunct to other lipid-lowering treatments (eg LDL apheresis) or if such treatments are unavailable.

Is also used to prevent cardiovascular events in adult patients who are thought to have a high risk for a first cardiovascular event, as an adjunct to correction of other risk factors.

Atorvastatin is a selective, competitive inhibitor of HMG-CoA reductase, the enzyme responsible for the conversion of 3-hydroxy-3-methyl-glutaryl-coenzyme A to mevalonate, a precursor of sterols, including cholesterol. The triglycerides and cholesterol in the liver are incorporated into very low density lipoproteins (VLDL) and released into the plasma for delivery to peripheral tissues. The low density lipoprotein (LDL) is formed from VLDL and is catabolized primarily through receptor high affinity to LDL (LDL receptor).

Atorvastatin lowers cholesterol levels and lipoprotein plasma inhibiting HMG-CoA reductase and then the biosynthesis of cholesterol in the liver and increase the number of LDL receptors on the surface of liver cells which uptake and catabolism of LDL. Atorvastatin reduces LDL production and the number of particles of LDL. H atorvastatin causes profound and sustained increase of LDL receptor activity, in combination with a beneficial change in the quality of the circulating particles of LDL. Atorvastatin effectively reduces LDL-C in patients with homozygous familial hypercholesterolemia, a group of patients who do not usually respond to lipid-lowering medicines.

Atorvastatin in a dose-response study, was shown to reduce the concentration of T-CHOL (30% - 46%), the LDL-CHOL (41% - 61%), apolipoprotein B (34% - 50%) and triglycerides (14% - 33%) while producing variable increases HDL-CHOL and apolipoprotein A1. These results are so consistent in patients with heterozygous familial hypercholesterolaemia, non-familial forms of hypercholesterolemia and mixed hyperlipidemia, including patients with noninsulin-dependent diabetes mellitus.

It has been found that the decrease of the values of total cholesterol, LDL-CHOL and apolipoprotein B reduces the risk of cardiovascular events and mortality thereof.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients (External Ambulatory) Patients.
* Male or female patients
* 18 to 99 years
* Patients with Hypercholesterolemia
* Patients with and without treatment with statin
* Patients enrolled in any of the study sites with acute cardiovascular event
* Patients discharged with study medication (Antorcin ®)
* Patients who have agreed and signed the consent form for the recording and processing of their personal data.

Exclusion Criteria:

* Patients under 18 and over 99 years.
* Women in pregnancy or lactation period
* Patients enrolled in any of the study sites for any reason other than an acute cardiovascular event
* Patients who discharged and take another statin drug formulation other than the study drug formulation (Antorcin ®)
* Patients who have not consented and signed the consent form for the recording and processing of their personal data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on atorvastatin treatment after hospitalization due to cardiovascular events
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change of lipids (LDL-C, HDL-C, T-CHOL)levels from baseline to the end of the studyCHOL) plasma blood Evaluation of atorvastatin (Antorcin) treatment per study subgroup | 0 months, 1-1,5 months, 4-4,5 months, 7-7,5 months
  The evaluation of atorvastatin treatment to all patients with cardiovascular events and separate the two subgroups (diabetes type II patients with metabolic syndrome) in order to achieve the level of lipids (LDL-C, HDL-C, T-CHOL) plasma blood
Change of LDL-C, HDL-C, T-CHOL from baseline to the end of the study by atorvastatin dosage scheme | 0 months, 1-1,5 months, 4-4,5 months, 7-7,5 months
  Achieving the level of lipids (LDL-C, HDL-C, T-CHOL) in blood plasma of patients in the atorvastatin dosage: those who received the 40 mg dose and those who received a dose of 80 mg

SECONDARY OUTCOMES:
Measurement of days without treatment - Patients' compliance | 0 months, 1-1,5 months, 4-4,5 months, 7-7,5 months
  The investigation of compliance to treatment (days without taking medication, changing the time of intake) and its correlation with the achievement of target lipid levels (LDL-C, HDL-C, T-CHOL) in blood plasma of the studied patients
Number of Adverse Events during study duration | 0 (baseline), 7-7,5 months
  Safety evaluation by adverse events reporting

OTHER OUTCOMES:
Changes in other than lipids hematological and biochemical parameters from baseline until the end of the study | 0, 1-1,5 months, 4-4,5 months, 7-7,5 months
  The reporting of hematological and biochemical tests where conducted at each hospital center, as part of their standard clinical practice
Number of participants per dyslipidemia categorization | 0 months (baseline)
  The determination of dyslipidemia class it belongs to each patient in order to assess the efficacy of atorvastatin administered.

CONTACTS AND LOCATIONS:
Overall Officials: Antonis Ziakas, Ass Professor, Principal Investigator — AHEPA hospital of Thessaloniki, Greece; Charalampos Karvounis, Professor, Principal Investigator — AHEPA hospital of Thessaloniki, Greece; Georgios Maligos, Registrat A, Principal Investigator — Papanikolaou hospital of Thessaloniki, Greece; Ioannis Kanonidis, Professor, Principal Investigator — Hippokration hospital of Thessaloniki, Greece; Dimitrios Psyropoulos, Director, Principal Investigator — Gennimatas hospital of Thessaloniki, Greece; Ioannis Vogiatzis, Director, Principal Investigator — Hospital of Veria, Greece; Pantelis Kligatsis, Director, Principal Investigator — Hospital of Florina, Greece; David Symeonidis, Director, Principal Investigator — Hospital of Kavala, Greece; Nikolaos Theodoridis, Director, Principal Investigator — Hospital of Drama, Greece; Stylianos Lampropoulos, Director, Principal Investigator — Hospital of Ptolemaida, Greece; Georgios Spyromitros, Director, Principal Investigator — Hospital of Katerini, Greece; Ioannis Tsounos, Director, Principal Investigator — Agios Pavlos hospital of Thessaloniki, Greece; Vlasis Pyrgakis, Director, Principal Investigator — George Gennimatas hospital of Athens, Greece; Andreas Tsellios, Registrat, Principal Investigator — NIMTS hospital of Athens, Greece; Ioannis Kalikazaros, Director, Principal Investigator — Hippokration hospital of Athens, Greece; Dimitrios Richter, Director, Principal Investigator — Euroclinic of Athens, Greece; Emmanouel Kallieris, Associate Director, Principal Investigator — Metropolitan hospital of Piraeus, Greece; Apostolos Katsivas, Director, Principal Investigator — Red Cross Hospital of Athens, Greece; Stefanos Foussas, Director, Principal Investigator — Tzannion hospital of Piraeus, Greece; Dimitrios Tziakas, Ass. Professor, Principal Investigator — University Hospital of Alexandroupolis, Greece; Konstantinos Papaioannou, Director, Principal Investigator — Hospital of Polygyros, Greece; Ioannis Styliadis, Director, Principal Investigator — Papageorgiou Hospital of Thessaloniki, Greece; Pantelis Makridis, Director, Principal Investigator — Hospital of Edessa, Greece; Panayotis Kyriakidis, Director, Principal Investigator — 424 military hospital of Thessaloniki, Greece; Georgios Karakostas, Director, Principal Investigator — Hospital of Kilkis, Greece; Vasilios Vasilikos, Ass Professor, Principal Investigator — Hippokration hospital of Thessaloniki, Greece; Sotirios Patsilinakos, Director, Principal Investigator — Konstantopoulio General Hospital of Athens; Dimitrios Sionis, Director, Principal Investigator — Sismanogleio General Hospital of Athens; Antonios Sideris, Director, Principal Investigator — Evagelismos General Hospital of Athens; Athanasios Manolis, Director, Principal Investigator — Asklepiion General Hospital of Voula; Chrysostomos Oikonomou, Director, Principal Investigator — Laikon General Hospital of Athens; Panagiotis Pentzeridis, Director, Principal Investigator — General State Hospital of Nikaia, Piraeus; Athanasios Pras, Director, Principal Investigator — General State Hospital of Chania, Crete; Alkiviadis Dermitzakis, Director, Principal Investigator — Venizeleio General State Hospital of Heraklion, Crete; Panagiotis Vardas, Professor, Principal Investigator — University Hospital of Heraklion, Crete; Dimitrios Alexopoulos, Professor, Principal Investigator — Rio University Hospital of Patras; Andreas Mazarakis, Director, Principal Investigator — Agios Andreas General State Hospital of Patras; Antonios Draganigos, Director, Principal Investigator — General State Hospital of Corfu; Filippos Tryposkiadis, Professor, Principal Investigator — University Hospital of Larisa, Thessaly; Spyridon Zombolos, Director, Principal Investigator — General State Hospital of Kalamata; Dimitrios Platogiannis, Director, Principal Investigator — General State Hospital of Trikala; Panagiotis Stasinos, Director, Principal Investigator — General State Hospital of Ierapetra, Crete; Nikitas Moschos, Director, Principal Investigator — General State Hospital of Rhodes; Chrysostomos Dilanas, Director, Principal Investigator — General State Hospital of Korinthos
Locations (17):
- Greece (17):
  - Rio University Hospital, Pátrai, Achaia
  - Euroclinic Private Hospital, Athens, Attica
  - Evagelismos General State Hospital, Athens, Attica
  - Gennimatas General State Hospital, Athens, Attica
  - Konstantopoulio General Hospital, Nea Ionia, Attica
  - General State Hospital, Polygyros, Chalkidiki
  - University Hospital, Heraklion, Crete
  - General State Hospital, Rhodes, Dodecanese
  - General State Hospital, Kalamata, Messinia
  - General State Hospital, Edesssa, Pella
  - 424 Military Hospital, Thessaloniki, Thessaloniki
  - Papageorgiou Hospital, Thessaloniki, Thessaloniki
  - University Hospital, Larissa, Thessaly
  - Hippokration General Hospital, Athens
  - Sismanogleio General State Hospital, Athens
  - General State Hospital, Nikaia Piraeus
  - Tzannion General State Hospital, Piraeus

REFERENCES:
- [Background] Thomas T, Ginsberg H. Development of apolipoprotein B antisense molecules as a therapy for hyperlipidemia. Curr Atheroscler Rep. 2010 Jan;12(1):58-65. doi: 10.1007/s11883-009-0078-7. PMID 20425272
- [Background] Benner JS, Glynn RJ, Mogun H, Neumann PJ, Weinstein MC, Avorn J. Long-term persistence in use of statin therapy in elderly patients. JAMA. 2002 Jul 24-31;288(4):455-61. doi: 10.1001/jama.288.4.455. PMID 12132975
- [Background] Jackevicius CA, Mamdani M, Tu JV. Adherence with statin therapy in elderly patients with and without acute coronary syndromes. JAMA. 2002 Jul 24-31;288(4):462-7. doi: 10.1001/jama.288.4.462. PMID 12132976
- [Background] Simons LA, Levis G, Simons J. Apparent discontinuation rates in patients prescribed lipid-lowering drugs. Med J Aust. 1996 Feb 19;164(4):208-11. doi: 10.5694/j.1326-5377.1996.tb94138.x. PMID 8604188
- [Background] Larsen J, Andersen M, Kragstrup J, Gram LF. High persistence of statin use in a Danish population: compliance study 1993-1998. Br J Clin Pharmacol. 2002 Apr;53(4):375-8. doi: 10.1046/j.1365-2125.2002.01563.x. PMID 11966668
- [Background] Frolkis JP, Pearce GL, Nambi V, Minor S, Sprecher DL. Statins do not meet expectations for lowering low-density lipoprotein cholesterol levels when used in clinical practice. Am J Med. 2002 Dec 1;113(8):625-9. doi: 10.1016/s0002-9343(02)01303-7. PMID 12505111
- [Background] Miettinen TA, Pyorala K, Olsson AG, Musliner TA, Cook TJ, Faergeman O, Berg K, Pedersen T, Kjekshus J. Cholesterol-lowering therapy in women and elderly patients with myocardial infarction or angina pectoris: findings from the Scandinavian Simvastatin Survival Study (4S). Circulation. 1997 Dec 16;96(12):4211-8. doi: 10.1161/01.cir.96.12.4211. PMID 9416884
- [Background] S Carter D Taylor. A Question of Choice: Compliance in Medicine Taking. Medicines Partnership 2003, www.medicines-partnership.org
- [Background] Seiki S, Frishman WH. Pharmacologic inhibition of squalene synthase and other downstream enzymes of the cholesterol synthesis pathway: a new therapeutic approach to treatment of hypercholesterolemia. Cardiol Rev. 2009 Mar-Apr;17(2):70-6. doi: 10.1097/CRD.0b013e3181885905. PMID 19367148
- [Background] Wei L, Wang J, Thompson P, Wong S, Struthers AD, MacDonald TM. Adherence to statin treatment and readmission of patients after myocardial infarction: a six year follow up study. Heart. 2002 Sep;88(3):229-33. doi: 10.1136/heart.88.3.229. PMID 12181210
- [Background] Heeschen C, Hamm CW, Laufs U, Snapinn S, Bohm M, White HD; Platelet Receptor Inhibition in Ischemic Syndrome Management (PRISM) Investigators. Withdrawal of statins increases event rates in patients with acute coronary syndromes. Circulation. 2002 Mar 26;105(12):1446-52. doi: 10.1161/01.cir.0000012530.68333.c8. PMID 11914253
- [Background] Thomas M, Mann J. Increased thrombotic vascular events after change of statin. Lancet. 1998 Dec 5;352(9143):1830-1. doi: 10.1016/S0140-6736(05)79893-7. No abstract available. PMID 9851392
- [Background] Guidelines of the Hellenic Society of Atherosclerosis for the diagnosis and treatment of dyslipidemia M. Elisaf, Ch. Pitsavos, E. Liberopoulos, V. Athyros Hellenic Journal of Atherosclerosis 2(3):163-168, 06/04/2011
- [Background] Davidson MH. Clinical significance of statin pleiotropic effects: hypotheses versus evidence. Circulation. 2005 May 10;111(18):2280-1. doi: 10.1161/01.CIR.0000167560.93138.E7. No abstract available. PMID 15883224